CLINICAL TRIAL: NCT04670419
Title: Morbidity and Mortality of Hepatitis E Virus Infections in Belgium 2010-2018
Brief Title: Morbidity and Mortality of Hepatitis E Virus Infections in Belgium
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Sciensano (Other Government); KU Leuven (Other)
Responsible Party: Principal Investigator, Thomas Vanwolleghem, Prof. Dr., University Hospital, Antwerp
Other Study IDs: 18/03/024
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hepatitis E
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples samples on which HEV serology (IgM and IgG), PCR and genotyping have been performed FFPE liver biopsy tissue blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HEV gt 3 clade abchijklm: patients infected with HEV gt 3 clade abchijklm
  Interventions: Other: Viral clade
- HEV gt 3 clade efg: patients infected with HEV gt 3 clade efg
  Interventions: Other: Viral clade

INTERVENTIONS:
Other: Viral clade — Disease outcomes are compared for patients infected with 2 different clades of a HEV gt 3 infection

SUMMARY:
Hepatitis E Virus (HEV) infections are emerging in the Western world with a predominance of HEV genotype (gt) 3. Except for age older than 50 years, male gender, chronic liver disease and immunosuppressed status, no correlators with clinical outcomes have been identified so far. With this study, we want to examine viral factors associated with the morbidity and mortality of HEV infections in Belgium as well as find correlators with clinical outcomes.

DETAILED DESCRIPTION:
1. Study objectives

   1.1. Primary objectives:

   To examine viral factors, such as gt, subtype and viral load, associated with the morbidity and mortality of HEV infections in Belgium.

   1.2. Secondary objectives:
   * To describe host factors associated with the morbidity and mortality of HEV infections in Belgium.
   * To find independent host and/or viral factors that are associated with the morbidity and mortality of HEV infections in Belgium.
2. Investigational plan

   2.1. General study design

   Retrospective cohort study.

   2.2. Study duration, enrollment and number of sites

   Subjects for which a serum sample is sent to the Belgian National Reference Center for Viral Hepatitis Sciensano to diagnose a HEV infection between January 2010 and June 2018.

   2.3. Study population

   All patients with a confirmed or possible HEV infection at Sciensano between January 2010 up to and included June 2018.

   2.3.1. Inclusion criteria:
   * HEV RNA positive AND/OR HEV immunoglobulin (Ig)M positive
   * Lab confirmation of the HEV infection performed at Sciensano
   * All ages will be included
   * Referring hospital in Belgium

   2.3.2. Exclusion criteria:
   * No confirmation of HEV serology AND/OR polymerase chain reaction (PCR) performed at Sciensano
   * Cases not diagnosed in Belgium
   * Cases without clinical outcome data
3. Study procedures

   Review of records. Re-evaluation of available liver biopsies by an expert liver pathologist (Prof. Tania Roskams, UZ Leuven).

   3.1. Data sources

   In Belgium, Sciensano acts as a National Reference Center (NRC) for viral hepatitis. Most of the documented HEV infections in Belgium are confirmed in Sciensano and samples on which HEV serology (IgM and IgG), PCR and genotyping have been performed are biobanked.

   3.2. Data collection

   A questionnaire will be sent to all treating physicians of patients with HEV infections in Belgium. If no response is received, a reminder will be sent by regular mail and later by e-mail. Different options will be offered to the treating physicians: to fill in the questionnaire, to complete the questionnaire by telephone with an investigator from Sciensano, to let the data to be collected at the center site by an investigator of Sciensano. Available liver biopsies from confirmed HEV cases will be retrieved from the pathology department of each center and re-evaluated by an expert liver pathologist.

   3.3. Variables collected

   Demographic data:

   Age and geographical origin. Date of symptom onset, date of diagnosis, date of loss to follow-up / death. Pregnancy at the time of diagnosis. Diabetes mellitus at the time of diagnosis. Immunocompromised status at the time of diagnosis. Known cirrhosis (fibroscan / biopsy / …), hematological or oncological disease. Other comorbidities. Blood transfusion history. Solid organ or stem cell transplantation preceding the HEV infection, type of organ and date. Renal function or renal replacement therapy. Infection in other family members. Use of alcohol and number of units per week. Use of illicit drugs. Travel abroad preceding the HEV infection and name of the country visited. Consumption of pork meat.

   Treatment data:

   Treatment with ribavirin. Treatment with other known/putative antiviral therapy. Reduction of immunosuppressive medication because of the HEV infection. Stop of immunosuppressive therapy because of HEV infection.

   Disease course and outcomes data:

   Acute hepatitis with complete recovery. Liver failure. Hospitalisation. Duration of hospitalisation in days. Admission to the intensive care unit. Duration of hospitalisation at the intensive care unit in days. Variceal bleeding. Bacterial peritonitis. Hepatic encephalopathy. Extrahepatic manifestations and type. Neurologic disease and type. Chronic HEV infection (as defined by HEV RNA positive for 3 months or more). Progression to cirrhosis as a consequence of HEV infection. Liver transplantation as a consequence of HEV infection and date of transplantation. Death and date of death. Death as a consequence of HEV infection. Total duration of symptoms in weeks.

   Biochemical data:

   HEV IgM, HEV IgG, HEV (quantitative) PCR, HEV genotype and subtype. HEV genotyping was performed by Sanger sequencing of a 348 base pair (between 2010 and 2016) or a 493 base pair (from 2017) region of ORF2. The obtained sequences were aligned against HEV reference genomes and submitted to HEVnet for genotype assignment (13). Presenting ALT, peak ALT, presenting AP, peak AP, presenting bilirubin, peak bilirubin, presenting INR, peak INR, presenting albumin, lowest albumin, presenting eGFR (CKD-EPI), lowest eGFR (CKD-EPI).

   Liver biopsy scoring:

   Histological grading and staging on H&E stained liver biopsy slides will be applied in a blinded manner. One expert liver pathologist, who is unaware of the infection status of the patient, will score the liver biopsies. The following parameters will be scored from 0-4 in a semi-quantitative manner: general architecture, lobular and portal inflammation, presence of immune cells and necrotic cells, presence of interfaces. Per patient, a global score will be assigned taken into account the spread, mean and mode of the different scored parameters.
4. Statistical analysis plan

The characteristics of patients will be analysed with the chi-square test for categorical variables and student t-test (Welch test if unequal variances or Wilcoxon Rank sum test when normality is not met) for the continuous variables. Numerical data are presented as the mean and standard deviation or 95% confidence interval, while categorical are expressed as counts and percentages.

The following independent viral variables are defined: HEV gt 3 clade type (abchijklm, efg and ra), viral load.

The following independent host variables are defined, given their known association with disease outcome or severity: alcohol consumption, diabetes, gender, age, cirrhosis and immunosuppression.

Differences between demographic factors, disease severity (expressed by laboratory data and histology) and disease outcomes (as defined by hospitalization status and duration, ICU stay, chronic infection, extrahepatic manifestations and death) will be analysed for the independent viral variables with an univariate analysis. Multivariable linear or logistic regression analysis will be performed with dependent variables that were found to be significantly associated with the independent variables in univariate analysis. Given the retrospective nature of the analysis, an upfront power calculation for the number of included patients for the investigated outcome is not possible. Statistical analyses are performed at a significance level of 5% using the statistical software R or SAS.

ELIGIBILITY:
Inclusion Criteria:

* HEV RNA positive AND/OR HEV immunoglobulin (Ig)M positive
* Lab confirmation of the HEV infection performed at Sciensano
* All ages will be included
* Referring hospital in Belgium

Exclusion Criteria:

* No confirmation of HEV serology AND/OR polymerase chain reaction (PCR) performed at Sciensano
* Cases not diagnosed in Belgium
* Cases without clinical outcome data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a confirmed or possible HEV infection at Sciensano between January 2010 up to and included June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
HEV viral factors associated with morbidity and mortality | observation period 2010-2018
  Viral factors, such as genotype, subtype and viral load, associated with the morbidity and mortality of HEV infections in Belgium

SECONDARY OUTCOMES:
Host factors associated with the morbidity and mortality of HEV infections in Belgium. | observation period 2010-2018
  Host factors, such as demographics and comorbidities

OTHER OUTCOMES:
independent host and/or viral factors associated with the morbidity and mortality of HEV infections in Belgium | observation period 2010-2018

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Vanwolleghem, MD PhD, Principal Investigator — University Hospital, Antwerp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peeters M, Schenk J, De Somer T, Roskams T, Locus T, Klamer S, Subissi L, Suin V, Delwaide J, Starkel P, De Maeght S, Willems P, Colle I, Van Hoof M, Van Acker J, Van Steenkiste C, Moreno C, Janssens F, Reynders M, Steverlynck M, Verlinden W, Lasser L, de Galocsy C, Geerts A, Maus J, Gallant M, Van Outryve S, Marot A, Reynaert H, Decaestecker J, Bottieau E, Schreiber J, Mulkay JP, de Goeij S, Salame M, Dooremont D, Dastis SN, Boes J, Nijs J, Beyls J, Hens N, Nevens F, Van Gucht S, Vanwolleghem T; Belgian Association for the Study of the Liver. Viral clade is associated with severity of symptomatic genotype 3 hepatitis E virus infections in Belgium, 2010-2018. J Hepatol. 2023 Jan;78(1):67-77. doi: 10.1016/j.jhep.2022.08.033. Epub 2022 Sep 6. PMID 36075495